CLINICAL TRIAL: NCT03859011
Title: Effectiveness and Cost-Effectiveness of Acupuncture for Chronic Neck Pain: A Pilot Randomized Controlled Trial
Brief Title: Acupuncture Relief for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 5 Element Institute (Other)
Collaborators: United States Naval Medical Center, Portsmouth (U.S. Federal Agency); Utica College (Other); RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NHJX.2021.0099
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Neck Pain, Posterior
Keywords: acupuncture; pain; neck pain
MeSH Terms: conditions — Neck Pain; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): After obtaining baseline data and questionnaires, patients will receive usual care (for example physical therapy, oral pain medication or neck injections), plus acupuncture 2X/week over 2 weeks, then once per week over 8 weeks (12 total treatments over 10 weeks), then no acupuncture between 10 weeks and 4 months. After treatment is completed, final measurement instruments are applied at 4 months. Questionnaires will be readministered at 2.5 and 4 months.
  Interventions: Other: Acupuncture
- "Usual" care (Placebo Comparator): After obtaining baseline data and questionnaires, patients will receive usual care (for example physical therapy, oral pain medication or ointments) for 4 months. Questionnaires will be readministered at 2.5 and 4 months.
  After the control phase the participants will continue usual care (for example physical therapy, oral pain medication or ointments), plus acupuncture 2X/week over 2 weeks, then once per week over 8 weeks (12 total treatments over 10 weeks, 6.5 months), then no acupuncture between 6.5 months and 8 months.
  Questionnaires will be readministered at 6.5 and 8 months.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Patients will have DBC Spring Ten acupuncture needles (manufactured in China) manually inserted bilaterally on five standardized acupuncture points according to the treatment points of GB20, BL10, BL11, SI3, BL62 at 6-8 mm depth for 20 minutes each using a tonification technique to elicit a de qi response.
  After those needles are removed, the number of additional needles and additional acupuncture points used will be chosen at the acupuncturist's discretion.

SUMMARY:
This study will assess the feasibility of measuring the effectiveness of "usual care" for chronic neck pain as defined in the protocol, compared with usual care plus acupuncture, for chronic neck pain. This study's hypothesis is that combining acupuncture with usual care will show a clinically relevant increase in the effectiveness of the integrated therapies, compared with usual care alone. This study will also assess the feasibility of measuring the cost-effectiveness of acupuncture for chronic neck pain. The hypothesis is that in economic evaluation terms, integrating acupuncture with usual care will not create significant overall costs, relative to the benefits which study patients obtain.

DETAILED DESCRIPTION:
Low back and neck pain accounts for the third-highest amount of U.S. healthcare spending, estimated at $87.6 billion annually. Moderate quality evidence already exists showing acupuncture's effectiveness for low back pain. Other than a few mostly foreign randomized controlled trials (RCTs) on acupuncture for neck pain, there are fewer quality studies on acupuncture's effectiveness for neck pain than for low back pain. The safety of acupuncture is well established. The risk of hematoma or infection due to acupuncture is lower than with venipuncture.

There is a lack of evidence on the cost-effectiveness relationship of this treatment strategy in the United States. A PubMed search found only three cost-effectiveness analyses of acupuncture for neck pain studies, all done abroad.

Since Medicare and several large private insurance companies still do not cover acupuncture for chronic neck pain, patient access to this therapy is significantly limited by out-of-pocket cost. A quality comparative effectiveness and cost-effectiveness study on acupuncture for chronic neck pain is needed from several perspectives. From the patient perspective, such a study would inform patients and providers in decision-making regarding integrating acupuncture in the care plan. From a third-party payer perspective, such a study would inform insurance companies whether it is cost-effective for them to cover acupuncture for this specific diagnosis. From a societal perspective, such a study would inform policy decision-makers whether acupuncture is a sound "investment" to better make resource allocation decisions for its citizens.

Pharmacological treatment of chronic pain has had safety issues. The CDC reports that over the past 10 years the average number of US drug-related deaths has exceeded 80,000 lives. The vast majority of these deaths have resulted from abuse and misuse of opioid drugs. The opioid crisis has added weight and urgency to finding safe and effective non-pharmacological therapies to treat chronic pain, including chronic neck pain.

1. The primary aim of this trial is to explore the feasibility of a large scale, multi-site comparative effectiveness trial of acupuncture plus "usual care" vs. usual care alone for reducing chronic neck pain.
2. The secondary aim of this trial is to explore the feasibility of cost-effectiveness evaluation of acupuncture for this condition from multiple perspectives.

The primary endpoint will be determined by comparing the mean change score on the Brief Pain Inventory (Short Form) from baseline (month 0) to the treatment completion (month 2.5), and 1.5 months after completion of the acupuncture treatment (month 4) between groups.

ELIGIBILITY:
Inclusion Criteria:

* Have Grade II neck pain with no signs or symptoms of major structural pathology but major interference with activities of daily living.
* Worst pain will be at least 4 out of 10 on the Brief Pain Inventory short form at the time of screening and a diagnosis of non-specific neck pain (axial and muscular neck pain, without radicular symptoms, is included) by a clinician based on history taking and physical examination, including any imaging examinations. Neck pain is defined as "pain, ache, or discomfort" in the area between the occiput and the third thoracic vertebra and between the medial borders of the scapulae.
* Have persistent or recurrent neck pain lasting longer than 3 months, and occurring at least once per week
* Have had at least one physician or emergency department visit for neck pain within the past 3 months AND be currently taking pain medication as prescribed, such as:

  * Acetaminophen
  * NSAIDS
  * Narcotics (≤ 30 Oral Morphine Equivalents (OME)
  * Robaxin (or equivalent)
* Be able to maintain a prone position for at least 20 minutes per the intervention methodology
* Be able to provide written informed consent.

Exclusion Criteria:

1. Have as their primary complaint radicular pain in the upper extremity with the distribution of a particular nerve root;
2. Report pain in another region that is more severe than the neck pain;
3. Have major hemorrhagic disease such as hemophilia;
4. Report a history of hypersensitive reaction to previous acupuncture treatment, metal allergy, or major skin hypersensitivities;

4. Have a history of cervical spine surgery, or be scheduled for cervical spine surgery, prior to enrollment in the study. However, subjects may be included if they have had a surgical consult but are not yet scheduled for surgery; 5. Be involved in known litigation related to neck pain; 6. Have head or neck cancer, or neck pain associated with ongoing radiation treatment to the head or neck; 7. Have a body mass index greater than 40; 8. Have a history of major psychiatric disability or cognitive instability; 9. Have a current or recent (within the past 6 months) history of alcoholism, or current or recent history of drug abuse, including abusing opioids or other controlled pain medication; 10. Have a known pregnancy; 11. Report a recent history of prior acupuncture treatment within the past three months. However, if the prior acupuncture treatment was for another region of the body and not systemic, such as auricular acupuncture, the exclusion period is within 6 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (Short Form) | Baseline though 8 months
  The Brief Pain Inventory (Short Form) will be used to measure neck pain at the time intervals noted in the Arms and Interventions section above. This validated instrument will be used to compare the effectiveness of the intervention between the Intervention arm and the Control arm.
  This instrument measures pain on an 11-point scale, from 0 to 10. A higher number indicates a worse outcome, and a lower number indicates a better outcome.
  Feasibility of study design and implementation will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: James Higgins, Captain MC USN ret., DO, Study Chair — Dept of Family Medicine, Naval Hospital Jacksonville
Locations (2):
- United States (2):
  - Naval Hospital Jacksonville, Jacksonville, Florida
  - 5 Element Institute, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] https://www.jointcommission.org/en-us/standards/national-performance-goals/pain-management
- [Background] Binder AI. Neck pain. BMJ Clin Evid. 2008 Aug 4;2008:1103. PMID 19445809
- [Background] van der Velde G, Yu H, Paulden M, Cote P, Varatharajan S, Shearer HM, Wong JJ, Randhawa K, Southerst D, Mior S, Sutton D, Jacobs C, Taylor-Vaisey A. Which interventions are cost-effective for the management of whiplash-associated and neck pain-associated disorders? A systematic review of the health economic literature by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Spine J. 2016 Dec;16(12):1582-1597. doi: 10.1016/j.spinee.2015.08.025. Epub 2015 Nov 26. PMID 26631759
- [Background] Willich SN, Reinhold T, Selim D, Jena S, Brinkhaus B, Witt CM. Cost-effectiveness of acupuncture treatment in patients with chronic neck pain. Pain. 2006 Nov;125(1-2):107-13. doi: 10.1016/j.pain.2006.06.006. Epub 2006 Jul 13. PMID 16842918
- [Background] Essex H, Parrott S, Atkin K, Ballard K, Bland M, Eldred J, Hewitt C, Hopton A, Keding A, Lansdown H, Richmond S, Tilbrook H, Torgerson D, Watt I, Wenham A, Woodman J, MacPherson H. An economic evaluation of Alexander Technique lessons or acupuncture sessions for patients with chronic neck pain: A randomized trial (ATLAS). PLoS One. 2017 Dec 6;12(12):e0178918. doi: 10.1371/journal.pone.0178918. eCollection 2017. PMID 29211741
- [Background] Vas J, Perea-Milla E, Mendez C, Sanchez Navarro C, Leon Rubio JM, Brioso M, Garcia Obrero I. Efficacy and safety of acupuncture for chronic uncomplicated neck pain: a randomised controlled study. Pain. 2006 Dec 15;126(1-3):245-55. doi: 10.1016/j.pain.2006.07.002. Epub 2006 Aug 23. PMID 16934402
- [Background] Liang Z, Zhu X, Yang X, Fu W, Lu A. Assessment of a traditional acupuncture therapy for chronic neck pain: a pilot randomised controlled study. Complement Ther Med. 2011 Jan;19 Suppl 1:S26-32. doi: 10.1016/j.ctim.2010.11.005. Epub 2010 Dec 23. PMID 21195292
- [Background] Irnich D, Behrens N, Molzen H, Konig A, Gleditsch J, Krauss M, Natalis M, Senn E, Beyer A, Schops P. Randomised trial of acupuncture compared with conventional massage and "sham" laser acupuncture for treatment of chronic neck pain. BMJ. 2001 Jun 30;322(7302):1574-8. doi: 10.1136/bmj.322.7302.1574. PMID 11431299
- [Background] Cho JH, Nam DH, Kim KT, Lee JH. Acupuncture with non-steroidal anti-inflammatory drugs (NSAIDs) versus acupuncture or NSAIDs alone for the treatment of chronic neck pain: an assessor-blinded randomised controlled pilot study. Acupunct Med. 2014 Feb;32(1):17-23. doi: 10.1136/acupmed-2013-010410. Epub 2013 Oct 30. PMID 24171895
- [Background] Cameron ID, Wang E, Sindhusake D. A randomized trial comparing acupuncture and simulated acupuncture for subacute and chronic whiplash. Spine (Phila Pa 1976). 2011 Dec 15;36(26):E1659-65. doi: 10.1097/BRS.0b013e31821bf674. PMID 21494196
- [Background] Aranha MF, Muller CE, Gaviao MB. Pain intensity and cervical range of motion in women with myofascial pain treated with acupuncture and electroacupuncture: a double-blinded, randomized clinical trial. Braz J Phys Ther. 2015 Jan-Feb;19(1):34-43. doi: 10.1590/bjpt-rbf.2014.0066. Epub 2014 Nov 28. PMID 25714602
- [Background] Dieleman JL, Baral R, Birger M, Bui AL, Bulchis A, Chapin A, Hamavid H, Horst C, Johnson EK, Joseph J, Lavado R, Lomsadze L, Reynolds A, Squires E, Campbell M, DeCenso B, Dicker D, Flaxman AD, Gabert R, Highfill T, Naghavi M, Nightingale N, Templin T, Tobias MI, Vos T, Murray CJ. US Spending on Personal Health Care and Public Health, 1996-2013. JAMA. 2016 Dec 27;316(24):2627-2646. doi: 10.1001/jama.2016.16885. PMID 28027366
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Health Sciences Policy; Committee on Pain Management and Regulatory Strategies to Address Prescription Opioid Abuse; Phillips JK, Ford MA, Bonnie RJ, editors. Pain Management and the Opioid Epidemic: Balancing Societal and Individual Benefits and Risks of Prescription Opioid Use. Washington (DC): National Academies Press (US); 2017 Jul 13. Available from http://www.ncbi.nlm.nih.gov/books/NBK458660/ PMID 29023083
- [Background] MacPherson H, Tilbrook H, Richmond S, Woodman J, Ballard K, Atkin K, Bland M, Eldred J, Essex H, Hewitt C, Hopton A, Keding A, Lansdown H, Parrott S, Torgerson D, Wenham A, Watt I. Alexander Technique Lessons or Acupuncture Sessions for Persons With Chronic Neck Pain: A Randomized Trial. Ann Intern Med. 2015 Nov 3;163(9):653-62. doi: 10.7326/M15-0667. PMID 26524571
- [Background] CDC National Center for Health Statistics Webpage: Provisional Drug Overdose Death Counts. 9/2025. https://www.cdc.gov/nchs/nvss/vsrr/drug-overdose-data.htm
- [Background] Tick H, Nielsen A, Pelletier KR, Bonakdar R, Simmons S, Glick R, Ratner E, Lemmon RL, Wayne P, Zador V; Pain Task Force of the Academic Consortium for Integrative Medicine and Health. Evidence-Based Nonpharmacologic Strategies for Comprehensive Pain Care: The Consortium Pain Task Force White Paper. Explore (NY). 2018 May-Jun;14(3):177-211. doi: 10.1016/j.explore.2018.02.001. Epub 2018 Mar 1. PMID 29735382
- [Background] Lee MS, Nielsen A, Kim TH, Ha IH, Harbin S, Wieland LS. Acupuncture for chronic neck pain (Protocol). Cochrane Database of Systematic Reviews, 2019.